CLINICAL TRIAL: NCT00406458
Title: A Phase 2 Repeat Dosing Clinical Trial of SB-509 in Subjects With Diabetic Neuropathy
Brief Title: Clinical Trial of SB-509 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-509-0601
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy
Keywords: Diabetic neuropathy; Diabetes Type I or II; Mild to moderate sensorimotor diabetic polyneuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Neuropathies | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-509 (Experimental): 60 mg SB-509 injected IM into lower limbs every 2 months
  Interventions: Drug: SB-509
- Normal Saline (Placebo Comparator): Normal saline injected IM into lower limbs every 2 months
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: SB-509 — 60 mg dose
  Arms: SB-509
Other: Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of the study is to study the clinical effects of the investigational drug, SB-509 versus placebo in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
SB-509 contains the gene (DNA-a kind of biological "blueprint") for a protein. When a researcher injects SB-509 into your legs, the drug enters the muscle and nerve cells around the injection site and causes these cells to make a protein. This protein causes your cells to increase production of another protein called vascular endothelial growth factor (VEGF), which may improve the structure and function of nerves. In addition, there are changes in the levels of 28 additional proteins in your cells. These proteins function to promote the growth of cells, are structures in cells, help synthesize products, and affect immune cells, and some have unknown functions. This increase in your own VEGF proteins may protect and repair the damaged nerves caused by diabetic neuropathy.

The study doctor will test SB-509 (60 mg) and placebo. Everyone in this study will receive intramuscular (IM-directly into the muscle) injections into both legs. This will happen 3 times over about 4 months. Two out of every 3 participants will receive SB-509 and 1 out of every 3 will receive placebo. You will not know, and the study doctor will not know, whether you will receive SB-509 or whether you will receive placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a clinical diagnosis of diabetes mellitus type I or II for at least 12 months prior to the study.
* Have received a diagnosis of mild to moderate sensorimotor diabetic neuropathy from a neurologist (a doctor who specializes in disorders of the nervous system) or endocrinologist (a doctor who specializes in diabetes). This type of neuropathy is a loss of sensation and muscle function that occurs in the legs and hands in a stocking and glove distribution. Subjects with diabetic neuropathy that results in loss of sensation or muscle function in only one nerve and results in loss of nerve function of the blood vessels and causes low blood pressure, will not be eligible.
* If female and of childbearing potential, agree to use a medically acceptable physical barrier method during the study.
* Have blood pressure < 140/90 mm Hg
* Body mass index (BMI) < 38 kg/m2

Key Exclusion Criteria:

Subjects with the following are NOT eligible to participate in this study:

* Have moderate to severe ischemic heart disease, any history of congestive heart failure, or have had a myocardial infarction (heart attack) within the previous 6 months.
* Have chronic foot or leg ulcers for >1 month, gangrene in the legs, or any previous amputation of the lower extremity.
* Have symptoms of intermittent claudication (or leg pain during exercise associated with peripheral artery disease) and/or an ankle brachial index (or a calculation of the difference between arm and leg blood pressures) of less than (<) 0.75.
* Have a history of cancer within the past 5 years (except for curable non-melanoma cancer of the skin, superficial bladder cancer in complete remission, or any other cancer that has been in complete remission for at least 5 years).
* Have colon polyps. If patients have a history of benign colonic polyps that have been removed, they must have evidence of a normal colonoscopy within the last 12 months.
* Require any drug that depresses patients' immune systems (such as methotrexate, cyclophosphamide, or cyclosporine) when they receive the study drug and for 30 days afterwards.
* Have a known disorder that affects patients' immune systems (such as HIV/AIDS, hepatitis B virus [HBV], hepatitis C virus [HCV], sarcoidosis, tuberculosis, rheumatoid arthritis, or autoimmune disorders).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for pain intensity (VASPI), Nerve Conduction Velocity (NCV), Total Neuropathy Score (TNS), Epidermal Nerve Fiber Density (ENFD) & Epidermal Nerve Fiber Density Regeneration (ENFDR) | One year

SECONDARY OUTCOMES:
Safety | One year

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - Coordinated Clinical Research, La Jolla, California
  - Advanced Medical Research, LLC, Lakewood, California
  - SF Clinical Research Center, San Francisco, California
  - Diablo Clinical Research, Walnut Creek, California
  - Bradenton Research Center, Bradenton, Florida
  - University of Miami, Diabetes Research Institute, Miami, Florida
  - Neurology Clinical Research, Sunrise, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Creighton Diabetes Center, Omaha, Nebraska
  - Upstate Clinical Research, Albany, New York
  - Peripheral Neuropathy Center, Weill Medical College of Cornell University, New York, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Nerve and Muscle Center of Texas, Houston, Texas
  - DGD Research, San Antonio, Texas
- Instituto Mexicano de Investigación Clinica, Mexico City, Col. Roma, Mexico

REFERENCES:
- See also: Sponsor website — http://www.sangamo.com